CLINICAL TRIAL: NCT00097877
Title: Comparison of the Effect on Glycemic Control of Biphasic Insulin Aspart 70/30 Versus Insulin Glargine in Combination With Metformin in Subjects With Type 2 Diabetes
Brief Title: Comparison of Biphasic Insulin Aspart 70/30 Versus Insulin Glargine in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-2191
Record Dates: First submitted 2004-11-30; First posted 2004-12-01 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart
Drug: insulin glargine

SUMMARY:
This trial is conducted in the United States of America (USA). The purpose of this study is to test whether Biphasic Insulin Aspart 70/30 twice a day with Metformin improves glycemic control vs. once daily Insulin Glargine with Metformin in subjects with Type 2 Diabetes who are inadequately controlled on basal insulin plus oral anti-diabetic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2005-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
HbA1c | After 24 weeks

SECONDARY OUTCOMES:
safety variables
8-point plasma glucose profile
other glycemic variables

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (64):
- United States (62):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Tuscaloosa, Alabama
  - Novo Nordisk Investigational Site, Vestavia Hills, Alabama
  - Novo Nordisk Investigational Site, Searcy, Arkansas
  - Novo Nordisk Investigational Site, Chula Vista, California
  - Novo Nordisk Investigational Site, Fullerton, California
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, New Britain, Connecticut
  - Novo Nordisk Investigational Site, Aventura, Florida
  - Novo Nordisk Investigational Site, Chiefland, Florida
  - Novo Nordisk Investigational Site, Fort Myers, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Boise, Idaho
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, New Albany, Indiana
  - Novo Nordisk Investigational Site, Des Moines, Iowa
  - Novo Nordisk Investigational Site, Overland Park, Kansas
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Baton Rouge, Louisiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Springfield, Massachusetts
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Cherry Hill, New Jersey
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Plainsboro, New Jersey
  - Novo Nordisk Investigational Site, New Hyde Park, New York
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, Syracuse, New York
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Kettering, Ohio
  - Novo Nordisk Investigational Site, Clinton, Oklahoma
  - Novo Nordisk Investigational Site, Tulsa, Oklahoma
  - Novo Nordisk Investigational Site, Eugene, Oregon
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Salem, Oregon
  - Novo Nordisk Investigational Site, Lancaster, Pennsylvania
  - Novo Nordisk Investigational Site, Melrose Park, Pennsylvania
  - Novo Nordisk Investigational Site, Norristown, Pennsylvania
  - Novo Nordisk Investigational Site, West Reading, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Lewisville, Texas
  - Novo Nordisk Investigational Site, Midland, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Ogden, Utah
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Warrenton, Virginia
  - Novo Nordisk Investigational Site, Bellevue, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Puerto Rico (2):
  - Novo Nordisk Investigational Site, Manatí
  - Novo Nordisk Investigational Site, Santurce

REFERENCES:
- [Result] Ligthelm RJ, Gylvin T, DeLuzio T, Raskin P. A comparison of twice-daily biphasic insulin aspart 70/30 and once-daily insulin glargine in persons with type 2 diabetes mellitus inadequately controlled on basal insulin and oral therapy: a randomized, open-label study. Endocr Pract. 2011 Jan-Feb;17(1):41-50. doi: 10.4158/EP10079.OR. PMID 20713345
- [Result] Oyer DS, Shepherd MD, Coulter FC, Bhargava A, Deluzio AJ, Chu PL, Trippe BS; Initiateplus Study Group. Efficacy and tolerability of self-titrated biphasic insulin aspart 70/30 in patients aged >65 years with type 2 diabetes: an exploratory post hoc subanalysis of the INITIATEplus trial. Clin Ther. 2011 Jul;33(7):874-83. doi: 10.1016/j.clinthera.2011.05.093. Epub 2011 Jul 8. PMID 21741089
- [Result] Trippe BS, Shepherd MD, Coulter FC, Bhargava A, Brett J, Chu PL, Oyer DS. Efficacy and safety of biphasic insulin aspart 70/30 in type 2 diabetes patients of different race or ethnicity (INITIATEplus trial). Curr Med Res Opin. 2012 Jul;28(7):1203-11. doi: 10.1185/03007995.2012.686444. Epub 2012 Jun 25. PMID 22509859
- [Derived] Bergenstal R, Lewin A, Bailey T, Chang D, Gylvin T, Roberts V; NovoLog Mix-vs.-Exenatide Study Group. Efficacy and safety of biphasic insulin aspart 70/30 versus exenatide in subjects with type 2 diabetes failing to achieve glycemic control with metformin and a sulfonylurea. Curr Med Res Opin. 2009 Jan;25(1):65-75. doi: 10.1185/03007990802597951. PMID 19210140
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com